CLINICAL TRIAL: NCT02621060
Title: Effect of the Administration of Chlorogenic Acid on Glucemic Control, Insulin Secretion and Insulin Sensitivity in Patients With Impaired Glucose Tolerance
Brief Title: Effect of Chlorogenic Acid on Patients With Impaired Glucose Tolerance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Esperanza Martínez-Abundis, Researcher Professor, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-ACG-271281-LYZ
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: Impaired Glucose Tolerance
Keywords: Chlorogenic acid; Control glucose; Insulin Secretion; Insulin Sensitivity
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance | interventions — Chlorogenic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 1200 mg dose per day, three capsules of 400 mg, times daily 1/ 2 hour before meals during 90 days.
  Interventions: Drug: Placebo
- Chlorogenic acid (Experimental): 1200 mg dose per day, three capsules of 400 mg, times daily 1/ 2 hour before meals during 90 days.
  Interventions: Drug: Chlorogenic acid

INTERVENTIONS:
Drug: Placebo — Placebo: 1200 mg per day for three months
  Other Names: Calcined magnesia
  Arms: Placebo
Drug: Chlorogenic acid — Chologenic acid: 1200 mg per day for three months
  Other Names: 3-O-Caffeoylquinic, acid Heriguard
  Arms: Chlorogenic acid

SUMMARY:
Chlorogenic acid has demonstrated promising effects in the treatment of glycemic control, obesity, dyslipidemia, insulin secretion, among others. The above mentioned findings show that Chlorogenic acid has an excellent potential for the control of glucose as well as insulin secretion and insulin sensitivity.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial was carried out in 30 patients with a diagnosis of impaired glucose tolerance in accordance with the American Diabetes Association criteria. The patients received 400 mg capsules of Chlorogenic acid or placebo, three times daily 1/ 2 hour before meals for 90 days. Before and after intervention the investigators evaluated: 2 hours plasma glucose, glycated hemoglobin (A1C), triglycerides, high-density lipoprotein, fasting glucose and blood pressure body weight, body mass index, waist circumference, total cholesterol, low-density lipoprotein, very-low-density lipoprotein, creatinine, aspartate transaminase and alanine transaminase.

Were calculated: Areas under the curve of glucose and insulin were calculated with de Trapezoidal formula. Total insulin secretion was evaluated with the Insulinogenic index and the insulin sensitivity was estimated using the Matsuda index.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 30.0-34.99 kg / m2.
* Diagnosis of IGT (OGTT Values between 140mg / dl and 199mg / dl.
* Written informed consent.
* Body weight stable over the last 3 months.
* Women in follicular phase of the menstrual cycle (days 3 to 8 of the cycle) at the time of laboratory tests.
* Women who are not contemplated get pregnant within the next 6 months.

Exclusion Criteria:

* Women pregnant or breastfeeding.
* Physical or mental disability that makes it impossible to perform the intervention.
* Diagnosis of Hypertension or heart failure.
* Smokers.
* Untreated thyroid disease.
* Consumption of oral agents or other medications or supplements with proven properties that modify the behavior of glucose and lipids (oral hypoglycemic agents, insulin, lipid-lowering).
* Diagnosis of liver disease or elevation twice of the upper normal value of liver enzymes.
* Diagnosis of renal disease or creatinine > 1.5 mg / dl.
* Diagnosis of Type 2 Diabetes Mellitus (T2DM) Fasting glucose ≥ 126 mg / dL and/or OGTT ≥ 200 mg / dL and/or A1C ≥ 6.5%.
* Total Cholesterol ≥ 280 mg/dL.
* Triglycerids ≥ 300 mg/dL.
* Known allergy to calcined magnesia or Chorogenic acid.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esperanza Martínez, PhD Science, Study Director — University of Guadalajara
Locations (1):
- Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] van Popele NM, Elizabeth Hak A, Mattace-Raso FU, Bots ML, van der Kuip DA, Reneman RS, Hoeks AP, Hofman A, Grobbee DE, Witteman JC. Impaired fasting glucose is associated with increased arterial stiffness in elderly people without diabetes mellitus: the Rotterdam Study. J Am Geriatr Soc. 2006 Mar;54(3):397-404. doi: 10.1111/j.1532-5415.2005.00614.x. PMID 16551305
- [Background] Shaw JE, Zimmet PZ, de Courten M, Dowse GK, Chitson P, Gareeboo H, Hemraj F, Fareed D, Tuomilehto J, Alberti KG. Impaired fasting glucose or impaired glucose tolerance. What best predicts future diabetes in Mauritius? Diabetes Care. 1999 Mar;22(3):399-402. doi: 10.2337/diacare.22.3.399. PMID 10097917
- [Background] Garber AJ, Handelsman Y, Einhorn D, Bergman DA, Bloomgarden ZT, Fonseca V, Garvey WT, Gavin JR 3rd, Grunberger G, Horton ES, Jellinger PS, Jones KL, Lebovitz H, Levy P, McGuire DK, Moghissi ES, Nesto RW. Diagnosis and management of prediabetes in the continuum of hyperglycemia: when do the risks of diabetes begin? A consensus statement from the American College of Endocrinology and the American Association of Clinical Endocrinologists. Endocr Pract. 2008 Oct;14(7):933-46. doi: 10.4158/EP.14.7.933. No abstract available. PMID 18996826
- [Background] Whiting DR, Guariguata L, Weil C, Shaw J. IDF diabetes atlas: global estimates of the prevalence of diabetes for 2011 and 2030. Diabetes Res Clin Pract. 2011 Dec;94(3):311-21. doi: 10.1016/j.diabres.2011.10.029. Epub 2011 Nov 12. PMID 22079683
- [Background] Garber AJ, Abrahamson MJ, Barzilay JI, Blonde L, Bloomgarden ZT, Bush MA, Dagogo-Jack S, Davidson MB, Einhorn D, Garvey WT, Grunberger G, Handelsman Y, Hirsch IB, Jellinger PS, McGill JB, Mechanick JI, Rosenblit PD, Umpierrez G, Davidson MH; American Association of Clinical Endocrinologists. AACE comprehensive diabetes management algorithm 2013. Endocr Pract. 2013 Mar-Apr;19(2):327-36. doi: 10.4158/endp.19.2.a38267720403k242. No abstract available. PMID 23598536
- [Background] Guerrero-Romero F, Rodriguez-Moran M, Perez-Fuentes R, Sanchez-Guillen MC, Gonzalez-Ortiz M, Martinez-Abundis E, Brito-Zurita O, Madero A, Figueroa B, Revilla-Monsalve C, Flores-Martinez SE, Islas-Andrade S, Rascon-Pacheco RA, Cruz M, Sanchez-Corona J. Prediabetes and its relationship with obesity in Mexican adults: The Mexican Diabetes Prevention (MexDiab) Study. Metab Syndr Relat Disord. 2008 Mar;6(1):15-23. doi: 10.1089/met.2007.0020. PMID 18370832
- [Background] American Diabetes Association. Standards of medical care in diabetes-2015 abridged for primary care providers. Clin Diabetes. 2015 Apr;33(2):97-111. doi: 10.2337/diaclin.33.2.97. No abstract available. PMID 25897193
- [Background] Adeney KL, Williams MA, Schiff MA, Qiu C, Sorensen TK. Coffee consumption and the risk of gestational diabetes mellitus. Acta Obstet Gynecol Scand. 2007;86(2):161-6. doi: 10.1080/00016340600994992. PMID 17364278
- [Background] McCarty MF. A chlorogenic acid-induced increase in GLP-1 production may mediate the impact of heavy coffee consumption on diabetes risk. Med Hypotheses. 2005;64(4):848-53. doi: 10.1016/j.mehy.2004.03.037. PMID 15694706
- [Background] Olthof MR, Hollman PC, Katan MB. Chlorogenic acid and caffeic acid are absorbed in humans. J Nutr. 2001 Jan;131(1):66-71. doi: 10.1093/jn/131.1.66. PMID 11208940
- [Background] Renouf M, Marmet C, Giuffrida F, Lepage M, Barron D, Beaumont M, Williamson G, Dionisi F. Dose-response plasma appearance of coffee chlorogenic and phenolic acids in adults. Mol Nutr Food Res. 2014 Feb;58(2):301-9. doi: 10.1002/mnfr.201300349. Epub 2013 Sep 4. PMID 24039147

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Chlorogenic Acid
Started | 15 | 15
Completed | 12 | 14
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Chlorogenic Acid | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Standard Deviation); unit: years] | 45 (9) | 43 (11) | 44 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 25
  Male | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  Mexico | 15 | 15 | 30
Body weight [Mean (Standard Deviation); unit: kg] — Body weight was evaluated through a bioimpedance digital scale and results are reported in kg with a decimal.
  kg | 81.3 (8) | 83.3 (9.8) | 82.3 (8.9)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 32.1 (2.5) | 32.6 (2.4) | 32.4 (2.4)
Waist circumference [Mean (Standard Deviation); unit: cm] — Waist circumference was measured with a flexible tape in them id point between the lowest rib and the iliac crest and is expressed in centimeters.
  cm | 103 (7) | 106 (10) | 105 (9)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of diastolic blood pressure (DBP). The value was expressed on mmHg
  mmHg | 120 (6) | 115 (11) | 117 (9)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of diastolic blood pressure (DBP). The value was expressed on mmHg.
  mmHg | 77 (6) | 77 (11) | 77 (9)
Fasting plasma glucose [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of fasting plasma glucose (FPG), was taken after an overnight fast and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
  mmol/L | 5.7 (0.4) | 5.7 (0.4) | 5.7 (0.4)
2-hour plasma glucose [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of 2-hour plasma glcuose (2-h PG), was taken two hours after the ingestion of the drink with 75 g dextrose and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
  mmol/L | 9.0 (0.5) | 8.8 (0.6) | 8.9 (0.6)
Glycated hemoglobin A1c [Mean (Standard Deviation); unit: Percent of glycated hemoglobin] | 5.6 (0.5) | 5.5 (0.3) | 5.5 (0.4)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of triglycerides (TG), was taken after an overnight fast and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
  mmol/L | 1.6 (0.7) | 1.6 (0.6) | 1.6 (0.7)
Total cholesterol [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of total cholesterol (TC) , was taken after an overnight fast and was evaluated by spectrophotometry method. The value was expressed on mmol/L.
  mmol/L | 4.9 (1.0) | 4.5 (0.6) | 4.7 (0.8)
High-density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of HDL-C, was taken after an overnight fast and was evaluated by colorimetric method. The value was expressed on mmol/L.
  mmol/L | 1.5 (0.4) | 1.7 (0.4) | 1.6 (0.4)
Low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for determining of LDL-C, was taken after an overnight fast and was calculated by Friedewald formula. The value was expressed on mmol/L.
  mmol/L | 2.6 (1.1) | 2.3 (1.0) | 2.5 (1.1)
Very low-density lipoprotein (VLDL) [Mean (Standard Deviation); unit: mmol/L] | 0.77 (0.36) | 0.72 (0.30) | 0.75 (0.40)
Glutamic oxaloacetic transaminase (GOT) [Mean (Standard Deviation); unit: IU/L] | 21.46 (14.72) | 18.16 (5.92) | 19.81 (11.15)
Glutamic pyruvic transaminase (GPT) [Mean (Standard Deviation); unit: IU/L] | 24.25 (8.51) | 20.93 (9.73) | 23.02 (10.60)
Creatinine [Mean (Standard Deviation); unit: mmol/L] | 0.05 (0.02) | 0.05 (0.02) | 0.05 (0.02)
Uric Acid [Mean (Standard Deviation); unit: mmol/L] | 0.32 (0.06) | 0.29 (0.05) | 0.3 (0.05)
Area under the curve of glucose (AUCG) [Mean (Standard Deviation); unit: mmol/L/min] — Area under the curve of glucose was obtained using the trapezoidal integration.
  mmol/L/min | 1139 (154) | 1119 (147) | 1129 (50)
Area under the curve of insulin (AUCI) [Mean (Standard Deviation); unit: pmol/L/min] — Area under the curve of insulin was obtained using the trapezoidal integration.
  pmol/L/min | 72,298 (24,627) | 76,993 (26,480) | 74,645 (25,238)
Total insulin secretion [Mean (Standard Deviation); unit: Unitless] — Total insulin secretion was calculated with the Insulinogenic index (Δ ABC insulin / Δ ABC glucose).
  Unitless | 0.58 (0.21) | 0.71 (0.25) | 0.65 (0.24)
First phase of insulin secretion [Mean (Standard Deviation); unit: Unitless] — Calculated by Stumvoll index [1283 + 1.829 · insulin 30 min (pmol/L) -138.7 · glucose 30 min (mmol/L) + 3.772 · insulin 0 min (pmol/L)]
  Unitless | 1248 (701) | 1331 (628) | 1289 (655)
Insulin sensitivity [Mean (Standard Deviation); unit: Unitless] — Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]
  Unitless | 2.17 (0.71) | 1.98 (0.88) | 2.07 (0.79)

OUTCOME MEASURES:

1. Primary Outcome: Fasting Plasma Glucose (FPG)
Description: Reflect the fasting glucose level after a 10- to 12-h overnight fast.
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Median (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
mmol/L | 5.8 (0.3) | 5.5 (0.4)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.05, Standard Deviation 2

2. Primary Outcome: 2 Hours Plasma Glucose (2-h PG)
Description: Subjects underwent a 2-h oral glucose tolerance test (2-h OGTT) by consuming 75-g of a dextrose load, and one sample was obtained 120 min after glucose administration.
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
mmol/L | 9.0 (0.8) | 8.5 (0.4)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.084, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Glycated Hemoglobin A1c (A1C)
Description: Shows what a person's average blood glucose level was for the 2 to 3 months before the test high-performance.
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: Percentage of A1C
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
Percentage of A1C | 5.8 (0.3) | 5.5 (0.4)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.755, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Total Insulin Secretion
Description: After intervention. Total insulin secretion was calculated with the Insulinogenic index (Δ ABC insulin / Δ ABC glucose).
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
Unitless | 0.55 (0.26) | 0.63 (0.25)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)

5. Primary Outcome: First Phase of Insulin Secretion
Description: After intervention with Stumvoll index
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
Unitless | 1281 (818) | 1133 (601)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.084, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Insulin Sensitivity
Description: After intervention Matsuda Index
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
Unitless | 2.43 (0.88) | 2.30 (1.23)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Area Under the Curve of Glucose
Description: Area under the curve of glucose was obtained using the trapezoidal integration.
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: mmol/l/min
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
mmol/l/min | 1187 (130) | 1145 (199)

8. Secondary Outcome: Area Under the Curve of Insulin
Description: Before and after intervention area under the curve of insulin
Time Frame: Week 12.
Measure: Mean (Standard Deviation); unit: pmol/L/min
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
pmol/L/min | 67,322 (31,531) | 72,857 (29,414)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.074, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Body Weight
Description: The weight was measured at baseline, week 4, week 8 and week 12 with a bioimpedance balance and the entered values reflect the weight at week 12
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
kg | 81.3 (7.9) | 80.8 (11.0)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.022, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Body Mass Index
Description: The Body Mass index was calculated at baseline and at week 12 with the Quetelet index and the entered values reflect the body mass index at week 12
Time Frame: Week 12.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
kg/m^2 | 32.0 (2.6) | 31.4 (2.7)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority; p = 0.022, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.05

11. Secondary Outcome: Waist Circumference (WC)
Description: Waist circumference was evaluated at baseline and at week 12 with a flexible tape and the entered values reflects the waist circumference measure at week 12
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
cm | 102 (5) | 104 (10)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority; p = 0.022, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.05

12. Secondary Outcome: Systolic Blood Pressure (SBP)
Description: The Systolic Blood Pressure was evaluated at baseline and week 12 with a digital sphygmomanometer and the entered values reflect the blood pressure at week 12
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
mmHg | 118 (9) | 113 (8)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.594, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Diastolic Blood Plessure (DBP)
Description: The Diastolic blood plessure was evaluated at baseline and week 12 with a digital sphygmomanometer and the entered values reflect the blood pressure at week 12
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
mmHg | 78 (7) | 74 (10)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.42, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Triglycerides (TG)
Description: The triglycerides were evaluated at baseline and week 12 with enzymatic-colorimetric techniques and the entered values reflect the triglycerides level at week 12
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
mmol/L | 1.7 (0.7) | 1.3 (0.5)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Total Cholesterol (TC)
Description: The total cholesterol was estimated by standardized techniques at baseline and week 12 and the entered values reflect the total cholesterol level at week 12
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
mmol/L | 5.3 (0.9) | 4.3 (0.5)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: High-density Lipoprotein Cholesterol (HDL-C)
Description: The HDL-C levels were evaluated at baseline and week 12 with enzymatic/colorimetric techniques and the entered values reflect the HDL-C level at week 12
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
mmol/L | 1.5 (0.3) | 1.8 (0.3)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.059, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Low-density Lipoprotein Cholesterol (LDL-C)
Description: The LDL-C levels were measured at baseline and at week 12 with standardized techniques and the entered values reflect the LDL-C levels at week 12
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
mmol/L | 2.7 (0.8) | 1.9 (0.5)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.049, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Very-low Density Lipoprotein (VLDL)
Description: The VLDL levels were measured at baseline and at week 12 with standardized techniques and the entered values reflect the c-LDL levels at week 12
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
mmol/L | 0.77 (0.32) | 0.61 (0.22)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Glutamic Pyruvic Transaminase (GPT)
Description: Before and after intervention by spectrophotometry
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
IU/L | 25.25 (13.46) | 22.64 (15.71)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.376, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Glutamic Oxaloacetic Transaminase (GOT)
Description: Before and after intervention by spectrophotometry
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
IU/L | 22.03 (10.91) | 17.79 (8.73)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.472, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Creatinine
Description: The creatinine levels were measured at baseline and at week 12 with standardized techniques and the entered values reflect the uric acid levels at week 12
Time Frame: Week 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
mmol/L | 0.06 (0.04) | 0.06 (0.02)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.774, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Uric Acid
Description: The uric acid levels were measured at baseline and at week 12 with standardized techniques and the entered values reflect the creatinina levels at week 12.
Time Frame: Week 12.
Population: 3 and 1 subjects dropout in the placebo and chlorogenic acid group respectively.
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Placebo | Chlorogenic Acid
Number analyzed (Participants) | 12 | 14
mmol/l | 0.34 (0.06) | 0.30 (0.09)
Statistical Analysis 1: Comparison: Chlorogenic Acid; Test type: Superiority or Other; p = 0.637, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected thoughtout the 90 days of the study
Arm/Group | Placebo | Chlorogenic Acid
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/15 | 2/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | Chlorogenic Acid (N=15)
Diarrea (Gastrointestinal disorders) | 3 | 1
Headacha (Nervous system disorders) | 0 | 2
polyuria (Renal and urinary disorders) | 2 | 1
abdominal pain (Gastrointestinal disorders) | 1 | 1
abdominal distention (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No